CLINICAL TRIAL: NCT06611163
Title: A Phase 3, Randomized, Double-blind, Placebo Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Subcutaneous Tildrakizumab in Subjects With Moderate to Severe Genital Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Tildrakizumab in Subjects With Moderate to Severe Genital Psoriasis.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TILD-24-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Moderate to Severe Genital Psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tildrakizumab 100 mg (Experimental)
  Interventions: Drug: Tildrakizumab 100 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Tildrakizumab 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Tildrakizumab 100 mg — Tildrakizumab 100 mg SC injection on Day 1, Week 4 and every 12 weeks thereafter
Drug: Placebo — Placebo SC injection at Day 1 and Week 4
  Arms: Placebo

SUMMARY:
Phase 3 study to evaluate the efficacy and safety of subcutaneous tildrakizumab in subjects with moderate to severe genital psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the trial, willingness and ability to comply with the protocol, and provide written informed consent in accordance with institutional and regulatory guidelines
2. Age ≥ 18 years of age at the time of signing consent
3. Diagnosis of moderate to severe psoriasis of the genital area at Screening and baseline defined as modified sPGA-G score of ≥3.
4. Presence of non-genital plaque psoriasis (BSA ≥1%) at both Screening and Baseline.
5. Presence of psoriasis of the genital area that is inadequately controlled with topical therapy or the subject is intolerant to topical therapy
6. Negative evaluation for TB within 4 weeks before initiating IMP, defined as a negative QuantiFERON test. Subjects with a positive QuantiFERON test or 2 successive indeterminate

QuantiFERON tests are allowed if they have all of the following:

* no history of active tuberculosis (TB) or symptoms of TB,
* a posteroanterior chest radiograph (with associated report available at the site) performed within 3 months of Screening with no evidence of active TB ( or of any other pulmonary infectious diseases),
* if prior latent TB infection, must have history of adequate prophylaxis (per local standard of care),
* if presence of latent TB is established, then treatment according to local country guidelines must have been followed for 4 weeks, prior to dosing in the study at Visit 2-Week 0.

A maximum of 2 QuantiFERON tests of no more than 3 weeks apart are allowed. A re-test is only permitted if the first is indeterminate; the result of the second test will then be used

Exclusion Criteria:

1. Predominantly non-plaque forms of psoriasis specifically erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new-onset guttate psoriasis.
2. Planned surgical intervention between Baseline and the Week 16 evaluation for a pre-treatment condition.
3. Active infection or history of infections as follows:

   * any active infection (bacterial, fungal or viral) for which systemic anti-infectives were used within 28 days prior to first investigational medicinal product (IMP) dose, with the last dose having been received within 7 days of Screening,
   * a serious infection, defined as requiring hospitalization or intravenous (IV) anti-infectives within 8 weeks prior to the first IMP dose, with the last dose having been received within 7 days of Screening,
   * recurrent or chronic infections, e.g., chronic pyelonephritis, chronic osteomyelitis, bronchiectasis, or other active infection that, in the opinion of the Investigator, might cause participation in this study to be detrimental to the subject.
4. Any concurrent medical condition or uncontrolled, clinically significant systemic disease ( e.g., renal failure, heart failure, hypertension, liver disease, diabetes, or anemia) that, in the opinion of the Investigator, could jeopardize subject safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with modified sPGA-G score of clear (0) or almost clear (1) with at-least a 2-point reduction from baseline | Week 16
  sPGA-G scale is a 6-point numerical scale that ranges from 0 (clear) to 5 (very severe)

SECONDARY OUTCOMES:
Proportion of subjects, with a baseline score of ≥ 4, who achieve at-least 4-point improvement in weekly average genital psoriasis itch numerical rating scale [GPI-NRS] within the GPSS for subjects | Week 16
  The GPI-NRS is a self-reported measure where participants will assess their psoriasis symptoms in the genital area and select a number on a scale of 0-10, where 0 represents no itch, and 10 represents the worst imaginable itch.
Mean change from baseline in the affected Body Surface Area (BSA) | Week 16
  The BSA will be measured using the palm method where the palm of the subject's hand (including the palmar aspect of the fingers) represents 1 % of the BSA. The affected areas are then calculated by their size compared to the subject's palm.
Change from baseline in genital psoriasis symptoms scale [GPSS] total score and individual items scores | Week 16
  The GPSS contains eight items regarding genital psoriasis symptoms. The items separately address itch, pain, discomfort, stinging, burning, redness, scaling, and cracking on an 11-point scale where 0 represents ''no symptom'' and 10 represents ''worst symptom imaginable".
  Each of the eight items are scored separately; in addition, a total score ranging from 0 (no genital psoriasis symptoms) to 80 (worst imaginable genital psoriasis symptoms) is reported.
Proportion of subjects with psoriasis area and severity index [PASI] 75 response | Week 16
  The PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no psoriasis on the body) to 72 (the most severe case of psoriasis).
Proportion of subjects with PASI 90 response | Week 16
  The PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no psoriasis on the body) to 72 (the most severe case of psoriasis).
Proportion of subjects with PASI 100 response, in subjects with BSA <10% | Week 16
  The PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no psoriasis on the body) to 72 (the most severe case of psoriasis).

CONTACTS AND LOCATIONS:
Locations (62):
- United States (38):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Smary Cures Clinical Research, Anaheim, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - T. Joseph Raoof MD, Inc./Encino Research Center, Encino, California
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - LA Universal Research Center Inc, Suite 1, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Therapeutics Clinical Research, San Diego, California
  - Dermatology Institute and Skin Care Center, Inc. DBA Clinical Science Institute, Santa Monica, California
  - Paradigm Clinical Research, Wheat Ridge, Colorado
  - Coral Gables Dermatology & Aesthetics, Coral Gables, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Homestead Associates in Research Inc, Homestead, Florida
  - Genomics Medical Research, Miami, Florida
  - Med-Care Research, Miami, Florida
  - Dermatology Affiliates Research Institute, LLC, Atlanta, Georgia
  - Mcintosh Clinic, PC, Thomasville, Georgia
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Oakland Hills Dermatology PC, Auburn Hills, Michigan
  - The Derm Institute of West Michigan, Caledonia, Michigan
  - Skin Specialists, PC, Omaha, Nebraska
  - Forest Hills Dermatology, Kew Gardens, New York
  - Equity Medical, New York, New York
  - The Moses H. Cone Memorial Hospital Operating Corporation, Greensboro, North Carolina
  - Hickory Dermatology Research Center, LLC, Hickory, North Carolina
  - Javara Inc/ Tryon Medical Partners, PLLC, Matthews, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Indiana Clinical Trials Center Optima Research Boardman, Boardman, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Advanced Research Experts, Nashville, Tennessee
  - Arlington Research Center, inc., Arlington, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
  - James Song, MD (James Song), Bellevue, Washington
- Bulgaria (5):
  - MC Medconsult-Lovech, Lovech
  - Medconsult Pleven, Pleven
  - Medical Centre Regina Life Clinic, Sofia
  - UMHAT Tsaritsa Yoanna-ISUL, Sofia
  - Diagnostic Consulatative Center, Sofia
- Georgia (5):
  - JSC Curatio, Tbilisi
  - New Vision Univestiry Hospital, Tbilisi
  - Aversi Clinic, Tbilisi
  - David Abuladze Clinic (DAC), Tbilisi
  - Raymann, Tbilisi
- Hungary (2):
  - University of Debrecen Dept of Dermatology, Debrecen, Hajdú-Bihar
  - Allergo-Derm Bakos Kft, Baross U 20.
- Poland (12):
  - Niepubliczny Zakladu Opieki Zdrowotnej MultiMedica s.c., Wroclaw, Lower Silesian Voivodeship
  - Luxderm Specjalistyczny Gabinet Dermatologiczny, Lublin, Lubslskie
  - Centrum Medyczne \All-Med\ spolka komandytowa, Krakow, Malopolska
  - Uniwersytecki Szpital Kliniczny, Klinika Dermatologii, Rzeszw, Podkarpackie Voivodeship
  - "Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Sp. z o.o", Malbork, Warmian-Masurian Voivodeship
  - Zdrowie Osteo-Medic s.c., Bialystok-Podlaskie
  - Care Access Gdansk, Gdansk
  - Care Access Holsamed Katowice, Katowice
  - Lidia Rajzer-Specjalistyczny Gabinet Dermatologiczno-Kosmetyczny, Krakow
  - Clinical Best Solution Sp. z o.o Sp. k. w Lublinie, Lublin
  - Clinical Best Solutions SP. Z.O.O. SP.K., Warsaw
  - Klinika Ambroziak, Warszswa